CLINICAL TRIAL: NCT00560482
Title: Phase II Randomized Double Blind Placebo-Controlled Study to Determine the Efficacy of ABR-215050 in Asymptomatic Patients With Metastatic Castrate-Resistant Prostate Cancer
Brief Title: Efficacy Study of ABR-215050 to Treat Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Active Biotech AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07TASQ08; EudraCT No: 2007-003470-26
Record Dates: First submitted 2007-11-15; First posted 2007-11-19 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Prostate Cancer
Keywords: prostate; cancer; prostatic cancer; castrate-resistant prostate cancer (CRPC)
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — tasquinimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: ABR-215050, tasquinimod
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABR-215050, tasquinimod — Gelatin capsules containing 0.25mg, 0.50mg, 1.0mg ABR-215050; 0.25mg/day taken orally once daily for 2 weeks, 0.50mg/day taken orally once daily for 2 weeks (dose-titration), and 1.0 mg/day taken once daily for 5 months (+6 months continuation)
  Arms: A
Drug: Placebo — Identical appearing gelatin capsules containing placebo
  Arms: B

SUMMARY:
To investigate ABR-215050 as a possible treatment for prostate cancer.

DETAILED DESCRIPTION:
For asymptomatic patients with Castrate-Resistant Prostate Cancer (CRPC), a "window of opportunity" is present. During this "window of opportunity" an intervention with little or no toxicity and the potential for extending the "symptom-free" period would be of great value to keep metastatic patients in an asymptomatic stage and thus delay the introduction of chemotherapy. The purpose of this study is to evaluate the safety and efficacy of ABR-215050 as an interventional agent for this role.

Overall survival for patients participating in study 07TASQ08 will be evaluated retrospectively using a separate study protocol 11TASQ11.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed diagnosis of adenocarcinoma of the prostate
* Asymptomatic metastatic CRPC (VAS pain score less than or equal to 3). The patient may take non-opioid analgesics for non-cancer pain discomfort
* Evidence of metastatic disease from CT or Bone scan
* Evidence of progressive disease after castration levels of testosterone have been achieved defined by any of the following criteria:

  * Increased serum prostate-specific antigen (PSA) levels (Confirmed by 3 consecutive PSA measurements within 1 year with at least 14 days between each measurement)
  * Progression of bidimensionally measurable soft tissue (nodal) metastasis: (CT scan or MRI)
  * Progression of bone disease: (New bone lesions by bone scan within the past 12 weeks)
* Castrate levels of serum testosterone (less than or equal to 50 ng/dL or 1.7 nmol/L. Testosterone levels will not be required for patients who have had bilateral orchiectomy)
* Karnofsky score 70-100
* Laboratory values as follows:

  * Hb greater than or equal to 90g/L (greater than or equal to 9g/dL)
  * Serum creatinine less than or equal to 1.5 x upper limit of normal (ULN)
  * Total bilirubin less than or equal to 1.5 x ULN
  * AST (SGOT) / ALT (SGPT) less than or equal to 2.5 x ULN
  * Serum amylase less than or equal to ULN. (If serum amylase is greater than ULN, pancreatic amylase and serum lipase should be analyzed. If both pancreatic amylase and serum lipase is greater than ULN, exclude patient)
* Patient if sexually active with partner of child bearing potential will agree to use adequate contraceptive methods (barrier contraceptive with spermicide or vasectomy) while on study drug
* No evidence (greater than or equal to 5 years) of prior malignancies (except successfully treated basal cell, squamous cell carcinoma of the skin)
* Ability to administer and retain oral medication
* Able to adhere to the study visit schedule and other protocol requirements

Exclusion criteria:

* Prior cytotoxic chemotherapy within 3 years
* Previous anti-cancer therapy using biologics or vaccines within the last 6 months. Previous treatment with bevacizumab is not allowed.
* Any treatment modalities, involving radiation and surgery, not discontinued at least 4 weeks prior to treatment in this study
* Myocardial infarction or any acute coronary syndrome within one year or current uncontrolled arrhythmias, symptomatic uncontrolled congestive heart failure, unstable angina pectoris, uncontrolled hypertension
* History of pancreatitis
* Any condition, including the presence of laboratory abnormalities, which confounds the ability to interpret data from the study or places the patient at unacceptable risk if he participates in the study
* Concurrent use of other anti-cancer agents or treatments [a stable dose of LHRH agonists, bicalutamide (e.g. Casodex) and/or other antiandrogens is allowed]
* Known brain metastases
* Simultaneous participation in any other study involving investigational drugs or having participated in a study less than 4 weeks prior to start of study treatment
* Concomitant systemic treatment with warfarin and/or corticosteroids corresponding to a prednisolone dose above 5 mg/day
* Exposure to ketoconazole or other strong CYP3A4 inhibitors or inducers intravenously or orally within 14 days prior to inclusion
* Known positive serology for HIV (patients with known history of HIV will be excluded because of potential for unforeseen toxicity and morbidity in an immunocompromised host)
* Chronic hepatitis with advanced, decompensated hepatic disease or cirrhosis of the liver or history of a chronic virus hepatitis or known viral hepatitis carrier (patients recovered from hepatitis will be allowed to enter the study)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2007-12; Primary Completion 2010-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Disease progression, defined as onset of tumor-related cancer pain, measurable disease progression, bone metastases or other non-target lesions, need for radiotherapy or surgery for pathological fracture or spinal cord compression | 3 months, 6 months; continuation phase every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Goran Forsberg, Assoc. Prof., Study Director — Active Biotech AB; Roberto Pili, MD, Principal Investigator — Roswell Park Cancer Institute, Buffalo, New York
Locations (65):
- United States (54):
  - Alaska Clinical Research Center LLC, Anchorage, Alaska
  - Southern California Permanente Medical Group, Anaheim, California
  - Southern California Permanente Medical Group, Baldwin Park, California
  - Southern California Permanente Medical Group, Bellflower, California
  - Pacific Clinical Center, Beverly Hills, California
  - South County Hematology/Oncology, Chula Vista, California
  - Southern California Permanente Medical Group, Fontana, California
  - Southern California Permanente Medical Group, Irvine, California
  - Cancer Center Oncology Medical Group, La Mesa, California
  - North County Oncology Medical Clinic, Inc., Oceanside, California
  - San Bernardino Urological Associates, San Bernardino, California
  - Urological Physicians of San Diego, Inc., San Diego, California
  - Southern California Permanente Medical Group, San Diego, California
  - Medical Oncology Associates - SD, San Diego, California
  - Sharp Memorial Hospital Investigational Pharmacy, San Diego, California
  - Sharp Rees-Stealy, San Diego, California
  - Pacific Clinical Research, Santa Monica, California
  - Agajanian Institute of Oncology and Hematology, Whittier, California
  - Porter Adventist Hospital, Denver, Colorado
  - Urology Associates, PC, Denver, Colorado
  - Diagnostic Professionals, Inc, Plantation, Florida
  - Southeastern Resarch Group, Inc., Tallahassee, Florida
  - Peachtree Hematology-Oncology Consultants, Atlanta, Georgia
  - St. Alphonsus Regional Medical Center, Boise, Idaho
  - North Idaho Urology, Coeur d'Alene, Idaho
  - Idaho Urologic Institute, PA, Meridian, Idaho
  - North Idaho Urology, Sandpoint, Idaho
  - University of Chicago, Chicago, Illinois
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Medical and Surgical Specialists, Galesburg, Illinois
  - OSF St Mary Medical Center, Galesburg, Illinois
  - Midwest Urology/RMD Clinical Research Institute, Melrose Park, Illinois
  - Johns Hopkins, Baltimore, Maryland
  - AdvanceMed Research, Lawrenceville, New Jersey
  - Urology Group of New Mexico, Albuquerque, New Mexico
  - Community Care Physicians, PC / The Urological Institute of Northeastern New York, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Beth Israel Medical Center, New York, New York
  - University Urological Associates, New York, New York
  - Staten Island Urological Research, PC, Staten Island, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Urological Associates, Raleigh, North Carolina
  - Urologic Consultants of SE PA, Bala-Cynwyd, Pennsylvania
  - Center for Urologic Care of the Main Line, Bryn Mawr, Pennsylvania
  - Urological Associates of Lancaster, Lancaster, Pennsylvania
  - University of Pittsburgh Physicians, Department of Urology, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - M.D. Anderson Cancer Center, Houston, Texas
  - Virginia Oncology Associates, Hampton, Virginia
  - Virginia Oncology Associates, Newport News, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Seattle Urology Research Center, Burien, Washington
  - Roger D. Fincher, M.D., P.S., Spokane, Washington
- Canada (8):
  - Andreou Research, Surrey, British Columbia
  - Surrey Memorial Hospital, Surrey, British Columbia
  - Guelph General Hospital, Guelph, Ontario
  - Guelph Nuclear Imaging, Guelph, Ontario
  - Guelph Urology Associates, Guelph, Ontario
  - Office of Dr. Bernard Goldfarb, North Bay, Ontario
  - 2150935 Ontario Inc., Owen Sound, Ontario
  - 3030 Lawrence Ave East, Scarborough Village, Ontario
- Sweden (3):
  - Institute of Clinical Sciences, Dept. of Urology / Sahlgrenska University Hospital, Gothenburg
  - University Hospital, Department of Urology, Malmo
  - Dept. of Urology, Akademiska Sjukhuset, Uppsala

REFERENCES:
- [Result] Pili R, Haggman M, Stadler WM, Gingrich JR, Assikis VJ, Bjork A, Nordle O, Forsberg G, Carducci MA, Armstrong AJ. Phase II randomized, double-blind, placebo-controlled study of tasquinimod in men with minimally symptomatic metastatic castrate-resistant prostate cancer. J Clin Oncol. 2011 Oct 20;29(30):4022-8. doi: 10.1200/JCO.2011.35.6295. Epub 2011 Sep 19. PMID 21931019
- [Result] Armstrong AJ, Haggman M, Stadler WM, Gingrich JR, Assikis V, Polikoff J, Damber JE, Belkoff L, Nordle O, Forsberg G, Carducci MA, Pili R. Long-term survival and biomarker correlates of tasquinimod efficacy in a multicenter randomized study of men with minimally symptomatic metastatic castration-resistant prostate cancer. Clin Cancer Res. 2013 Dec 15;19(24):6891-901. doi: 10.1158/1078-0432.CCR-13-1581. Epub 2013 Nov 19. PMID 24255071